CLINICAL TRIAL: NCT06532513
Title: Examination of the Effects of Family-Centered Goal-Oriented Physiotherapy and Rehabilitation Application on Body Functions, Activity, Participation and Quality of Life in Severely Affected Children With Dyskinetic Cerebral Palsy
Brief Title: Family-Centered Physiotherapy in Dyskinetic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mintaze Kerem Gunel, pt, PhD, prof., Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/13-07 (KA-22031)
Record Dates: First submitted 2024-07-22; First posted 2024-08-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy, Dyskinetic
Keywords: Dyskinetic Cerebral Palsy; Family-Centered Care; Physiotherapy; Rehabilitation; Body Functions; Activities of Daily Living; Participation; Quality of Life; Children's Health; Motor Skills Disorders
MeSH Terms: conditions — Cerebral Palsy; Motor Skills Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Family-Centered Goal-Oriented Physiotherapy and Rehabilitation Application (Experimental): Participants in this group will receive routine physiotherapy and rehabilitation for 10 weeks, along with an additional 1-hour training for family centered goal-oriented physiotherapy and rehabilitation practices. Families will be instructed to perform these practices at home for 1 h every day.
  Interventions: Other: Family-Centered Goal-Oriented Physiotherapy and Rehabilitation Application
- Control Group: Routine Physiotherapy and Rehabilitation Program (No Intervention): Participants in this group will undergo routine physiotherapy and rehabilitation for 10 weeks.

INTERVENTIONS:
Other: Family-Centered Goal-Oriented Physiotherapy and Rehabilitation Application — Family centered goal-oriented physiotherapy and rehabilitation applications aim to enhance the functional level of severely affected children with dyskinetic cerebral palsy children through individualized activities conducted by family members at home. The program focuses on specific goals determined collaboratively by the family, physiotherapists, and physician, with regular monitoring and assessments to track progress.
  Arms: Experimental Group: Family-Centered Goal-Oriented Physiotherapy and Rehabilitation Application

SUMMARY:
This study aimed to examine the impact of family centered, goal-oriented physiotherapy and rehabilitation on body function, activity, participation, and quality of life in severely affected children with dyskinetic cerebral palsy (DCP). The first assessment was conducted and recorded for all patients at the beginning of the study. Subsequently, the study group was taught family centered physiotherapy practices in addition to routine physiotherapy for 10 weeks to be performed at home. The control group only received routine physiotherapy. Weekly remote monitoring, regular meetings, and a second assessment at the 10th week were conducted. The study concluded with all face-to-face assessments.

According to the research protocol, the primary aim of this study was to evaluate the effectiveness of a 10-week family centered physiotherapy application. The goal of this intervention was to improve movement and posture, thereby enhancing daily activities and quality of life. The primary endpoint of the study was to determine the impact of family physiotherapy application taught to families during the 10-week education period.

This study was conducted at the Faculty of Physical Therapy and Rehabilitation, Hacettepe University. This study aimed to structure and define a family centered, goal-oriented, personalized physiotherapy, and rehabilitation application for the treatment of children with cerebral palsy. One of the significant objectives of this study was to examine the effects of this intervention within the framework of the International Classification of Functioning, Disability, and Health (ICF) on body function, activity, participation, and quality of life. The study protocol started with evaluations from patients after obtaining approval from the ethics committees.

The study will be completed within a follow-up period of four months without treatment, including the remote monitoring process. The results of this study aimed to provide valuable information about the effectiveness of family centered physiotherapy application in severely affected children with dyskinetic cerebral palsy.

DETAILED DESCRIPTION:
This study aimed to investigate the impact of family centered goal-directed physiotherapy and rehabilitation intervention on body function, activities, participation, and quality of life in children with severely affected dyskinetic cerebral palsy. Within this scope, an intervention program was designed to enhance children's functional performance in their daily life activities. The focal points of this research included pain, fatigue, sleep problems, and parental stress levels. The goal of this intervention was to improve children's movement and posture, increase their independence in daily life activities, and enhance their overall quality of life. This study aimed to assess the effectiveness of family centered interventions in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

1. Being in the age range of 5-18 years
2. Having a diagnosis of Dyskinetic Cerebral Palsy (DSP) confirmed by a pediatric neurologist
3. Being classified with a gross motor function level of IV-V using the Expanded and Revised Gross Motor Function Classification System (GMFCS E&R)
4. Having a Manual Ability Classification System (MACS) classification of manual ability level IV-V
5. Having a Communication Function Classification System (CFCS) communication function level of I-II-III
6. For volunteers participating through Zoom and Whatsapp applications, having computer literacy and these applications installed on their devices

e. Continuing routine physiotherapy and rehabilitation programs.

Exclusion Criteria:

1. Having difficulty understanding and following instructions
2. Having severe visual impairments
3. Having undergone orthopedic or brain surgery interventions in the last 12 months.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The Gross Motor Function Measure-88; The Gross Motor Function Measure-66 | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Gross Motor Function Measure-88 (GMFM-88) and its short form, the Gross Motor Function Measure-66( GMFM-66), assess gross motor function in children, especially those with cerebral palsy. KMFÖ-88 is widely used for comprehensive evaluations in clinical and research settings, whereas GMFM-66-66, a shorter version, focuses on activity measurement based on the International Classification of Functioning, Disability, and Health for Children and Youth (ICF-CY) to evaluate functional capacity in different positions and activities. A physiotherapist will conduct the assessment through clinical testing and video recordings will be independently evaluated by another researcher.

SECONDARY OUTCOMES:
Dyskinesia Impairment Scale | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Dyskinesia Impairment Scale (DIS) was used to assess the duration and amplitude of distonia and choreoathetosis in 12 body regions, including the eyes, mouth, neck, trunk, and extremities. It provides scores for each region during both action and rest, resulting in a total action score ranging from 0 to 192 and a total rest score ranging from 0 to 96 for both the subscales. The action and rest scores combine to create a total score between 0 and 288, representing the sum of the distonia and choreoathetosis subscales.
Dyskinesia Impairment Mobility Scale | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Dyskinesia Impairment Mobility Scale (DIMS) assesses dyskinesia in motorized wheelchair mobility performance. It has two subscales, Dyskinesia-Dystonia (DIMS-D) and Dyskinesia-Choreoathetosis (DIMS-CA), which use video-based protocols. Each subscale evaluated dyskinesia duration (time during mobility tasks) and amplitude (maximum Range of Motion (ROM) due to dyskinesia) in five motorized mobility tasks. The scores ranged from 0 to 4 for both factors. DIMS assesses overflow movements during mobility tasks and voluntary movements for wheelchair navigation, representing various body regions. The assessment covers the neck and proximal and distal parts of the right and left arms, excluding the feet. DIMS is excluded for assessing the feet due to minimal movement during wheelchair acceleration and braking.
Wong-Baker Faces Pain Rating Scale | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Wong-Baker FACES Pain Rating Scale was employed for pain assessment, particularly for patients aged 3 and above. This validated and recommended scale represents pain levels through facial expressions. The scale ranges from face 0, indicating no pain, to face 5, representing the possibility of the worst pain. The faces expressed increasing levels of pain intensity, with face 1 for mild pain, face 2 for moderate pain, face 3 for severe pain, and face 4 for very severe pain.
Dyskinetic Cerebral Palsy Functional Impact Scale | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  Dyskinetic Cerebral Palsy Functional Impact Scale (D-FIS) assesses the impact of dyskinesia on daily activities in children with DSP, featuring 18 items, including Pain and Fatigue, and 16 items on daily activities. Parent-proxy completion takes 10 minutes; D-FIS scores on the Impact Scale (0-72) and Priority Scale (1-4) evaluate dyskinesia impact and activity priority. Ratings consider unassisted functions and offer comprehensive evaluation. Higher scores suggest a greater dyskinesia impact, guiding intervention focus on priority areas for children and families.
Gross Motor Function Classification System | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Gross Motor Function Classification System (GMFCS) was used to assess gross motor function.
Manual Ability Classification System | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Manual Ability Classification System (MACS) was used to assess fine motor skills.
Communication Function Classification System | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Communication Function Classification System (CFCS) was used for assess communication function.
  The Communication Function Classification System (CFCS) is USED for ASSESSING communication function.
Eating and Drinking Classification System | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the interventione
  The Eating and Drinking Classification System (EDACS) was used for assess eating and drinking skills.
Visual Function Classification System | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Visual Function Classification System (VFCS) was used for assess visual function.
Goal Attainment Scale | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  To assess and measure the impact of individualized goal-oriented physiotherapy and rehabilitation programs on children with SP, the Goal Attainment Scale (GAS) was employed. To evaluate the effectiveness of the intervention, specific goals determined by the child, family, and experts were rated on a scale from -2 to 2, representing five levels of achievement. These goals are established through collaboration between the physiotherapist and family, and the attainment of these goals after the intervention is evaluated through discussions between the physiotherapist and family.
Life-Habits Questionnaire | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Life-Habits Questionnaire (Life-H) was used to assess the multidimensional aspects of children's participation. Life-H examines the participation of children with SP in various life activities under 12 subheadings, including participation in daily activities and social roles, providing both total and subsection scores. The daily activities include six subscales: "nutrition," "physical fitness," "personal care," "communication," "housing," and "mobility," while the social roles encompass "responsibilities," "interpersonal relationships," "social life," "education," "employment," and "leisure activities." Achievement scores range from 0 (failed or not completed) to 9 (performed without difficulty and assistance), varying based on the degree of difficulty and type of assistance required to accomplish a task. The Turkish version of Life-H has been demonstrated to be valid and reliable for assessing participation in children with SP.
European Child Environment Questionnaire | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The European Child Environment Questionnaire (ECEQ) will be used to assess environmental factors, considering that environmental factors can influence assessment outcomes when evaluating children using different assessment methods and recognizing the need for a comprehensive evaluation within the framework of the International Classification of Functioning, Disability, and Health (ICF). The ECEQ, consisting of 60 questions assessing conditions in the home, school, and community under three main subheadings: physical environment, social support, and attitudes, was designed to evaluate environmental factors in children with SP and determine their needs and accessibility. The scale is valid and reliable. Scoring is done on a scale of 0 (not necessary), 1 (necessary and mostly accessible), or 2 (necessary but mostly inaccessible) to determine the necessity and accessibility of needs.
Parental Stress Scale | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Parental Stress Scale (PSS) was used to assess parental stress (Appendix-11). It was utilized to evaluate the perceived parental stress levels of parents of children with SP participating in the study. The scale employs 18 items to measure parenting stress, considering the impact of children on the parental role and avoiding questions that could be confounded by general stress. Items are scored on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score, ranging from 18 to 90, was obtained by summing the sub-scores of the four main areas: rewards, loss of control, stressors, and satisfaction. Higher scores indicated higher levels of parenting stress. The psychometric properties of this scale have recently been shown to be adequate for families with chronic health conditions.
Cerebral Palsy Quality of Life Questionnaire Child and Teen Palsy Quality of Life Questionnaire Child&Teen | Time frame1: baseline, pre-intervention; Time frame 2: immediately after the intervention
  The Cerebral Palsy Quality of Life Questionnaire Child and Teen (CP QOL Child&Teen) will be utilized to assess the quality of life. It consists of two versions: one completed by the caregiver and another self-administered by the adolescent. The adolescents' self-administered questionnaire included six categories: family and friends, school, participation, communication, health, and special equipment, which were assessed under four subsections: general well-being and participation, communication and physical health, school situation, and social well-being. In addition, the caregiver questionnaire included two additional categories for evaluating services and family health. Respondents used a 9-point Likert scale to answer the questionnaire items based on the nature of the questions, marking a number from 1 to 9, indicating responses such as very unhappy, very important-not important at all, never sad-very sad, and no pain at all.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Günbey, PhD, Study Director — Hacettepe University; Eda Burç, MSc, Study Director — Hacettepe University
Locations (1):
- EDA BURÇ, Ankara, Hacettepe University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No